CLINICAL TRIAL: NCT03930498
Title: PD-1 Antibody Combined With Chemotherapy in High-risk Recurrent Nasopharyngeal Carcinoma: a Prospective, Open, Single-arm Phase II Clinical Trial
Brief Title: Programmed Death-1 (PD-1) Antibody Combined With Chemoradiotherapy in High-risk Recurrent Nasopharyngeal Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhao Chong, Prof., Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: High-risk rNPC-JS001
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: PD-1 antibody; Intensity-modulated Radiation Therapy; Chemotherapy; Efficacy; Adverse effects
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody plus chemoradiotherapy (Experimental)
  Interventions: Drug: PD-1 blocking antibody; Drug: Chemotherapy; Radiation: IMRT

INTERVENTIONS:
Drug: PD-1 blocking antibody — Toripalimab is an antibody targeting PD-1 developed by Shanghai Junshi Biosciences Co., Ltd.
  Other Names: JS001
Drug: Chemotherapy — Cisplatin and Gemcitabine
Radiation: IMRT — IMRT 60-66Gy, 1.8-2.0Gy/f/day

SUMMARY:
This is a a prospective, single-arm phase II clinical trial. The purpose of this study is to evaluate the efficacy and adverse effect of PD-1 antibody with chemotherapy in high-risk recurrent nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as local recurrence ± regional recurrence after ≥1 year of radical treatment;
* Not suitable for surgery;
* Newly histologic diagnosis of NPC (WHO II/III);
* Clinical stage rII-IVa (AJCC/UICC 8th);
* ECOG 0-1 point;
* PRANCIS score > 252 points;
* No treatment to rNPC, such as radiotherapy, chemotherapy, immunotherapy or biotherapy;
* No contraindications to immunotherapy or chemoradiotherapy;
* Adequate marrow function: WBC count ≥ 3×10E9/L, NE count ≥ 1.5×10E9/L, HGB ≥ 90g/L, PLT count ≥ 100×10E9/L;
* Adequate liver function: ALT/AST ≤ 2.5×ULN, TBIL ≤ 2.0×ULN;
* Adequate renal function: BUN/CRE ≤ 1.5×ULN or endogenous creatinine clearance ≥ 60ml/min (Cockcroft-Gault formula);
* Take effective contraceptions during and two months after treatment;
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* Have recurrence with local necrosis;
* Have ≥G3 late toxicities, except for skin, subcutaneous tissue or mucosa;
* Unexplained fever > 38.5 ℃, except for tumor fever;
* Treated with ≥ 5 days antibiotics one month before enrollment;
* Have active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy);
* Have a known history of human immunodeficiency virus (HIV), active Hepatitis B (HBV-DNA ≥10E3copiers/ml) or hepatitis C virus (HCV) antibody positive;
* Have previously treated with PD-1 antibody or other immunotherapy for PD-1/PD-L1 pathway;
* Have New York Heart Association (NYHA) class 3 or 4, unstable angina, myocardial -infarction within 1 year, or clinically meaningful arrhythmia that requires treatment;
* Have known allergy to large molecule protein products or any compound of study therapy;
* Pregnant or breastfeeding;
* Prior malignancy except adequately treated non-melanoma skin cancer, in situ cervical cancer, and papillary thyroid carcinoma;
* Have received a live vaccine within 30 days of planned start of study therapy Has psychiatric drug or substance abuse disorders that would interfere with cooperation with the requirements of the trial;
* Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  From date of recruitment to death

SECONDARY OUTCOMES:
Objective response rate | After 3 cycles of GP chemothrapy plus PD-1 antibody (each cycle is 21 days)
  Patient's short-term effect
Disease control rate | After 3 cycles of GP chemothrapy plus PD-1 antibody (each cycle is 21 days)
  Patient's short-term effect
Progression free survival | 2 years
  From date of recruitment to disease progression or death
Adverse effects | through study completion, an average of 3 months
  Evaluating with CTCAE v5.0
Quality of life: EuroQoL 5 dimension | through whole study, an average of 2 years
  Evaluating with questionnaire of EuroQoL 5 dimension, 5 level health state utility index (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, M.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Home Page of Sun Yat-sen University Cancer Center — http://www.sysucc.org.cn